CLINICAL TRIAL: NCT04252846
Title: A Prospective, Non-Interventional, Observational, Multicenter Study to Investigate Dosage, Effectiveness, and Safety of Perampanel When Used as First Adjunctive Therapy in the Routine Clinical Care of Subjects >=12 Years With Partial Onset Seizures With or Without Secondary Generalization or With Primary Generalized Tonic-Clonic Seizures Associated With Idiopathic Generalized Epilepsy
Brief Title: A Study to Investigate Dosage, Effectiveness, and Safety of Perampanel When Used as First Add-on Therapy in Participants >=12 Years With Partial Onset Seizures With or Without Secondary Generalization or With Primary Generalized Tonic-Clonic Seizures Associated With Idiopathic Generalized Epilepsy
Status: Completed | Type: Observational
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2007-M044-512
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-12

CONDITIONS: Idiopathic Generalized Epilepsy; Partial Onset Seizures; Generalised Tonic-Clonic Seizures
Keywords: Perampanel; Fycompa; Epilepsy; Seizures; Prospective
MeSH Terms: conditions — Epilepsy, Idiopathic Generalized; Epilepsy, Tonic-Clonic; Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perampanel: Participants with a diagnosis of epilepsy (POS with or without SG or PGTCS associated with IGE) will initiate treatment with perampanel as first adjunctive treatment as per the clinical judgment of the treating physician as part of routine clinical care. All participants will be observed prospectively for up to 12 months after initiation of perampanel treatment.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel oral tablets or oral suspension.
  Other Names: Fycompa

SUMMARY:
The primary purpose of this study is to assess the retention rate of perampanel as a reliable proxy for overall effectiveness and tolerability in participants aged at least 12 years who are prescribed perampanel (for partial onset seizures [POS] with or without secondary generalization [SG] or for primary generalized tonic-clonic seizures [PGTCS] associated with idiopathic generalized epilepsy [IGE] as first adjunctive to antiepileptic drug (AED) monotherapy as part of their routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of epilepsy
2. History of POS with or without SG or PGTCS associated with IGE
3. Documented POS with or without SG or PGTCS associated with IGE, within the past 12 months
4. Previously treated with 1 or 2 AEDs as monotherapy
5. At least 4 weeks' seizure diary data, or sufficient clinical detail to calculate baseline seizure frequency

Exclusion Criteria:

1. Episode(s) of status epilepticus within the past 6 months before Screening
2. Previously treated with 2 or more AEDs in combination (other than during cross-titration between AED monotherapies)
3. Previous or current use of perampanel

   Note: Retrospective inclusions will be allowed but only if the time between the initiation of perampanel treatment and the inclusion does not exceed 7 calendar days
4. Hypersensitivity to perampanel or any of the excipients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 300 participants with diagnosis of epilepsy (POS with or without SG or PGTCS associated with IGE)
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Retention Rate at Month 12 | Month 12
  Retention rate at 12 months is defined as the percentage of participants remaining on perampanel at 12 months.

SECONDARY OUTCOMES:
Retention Rate at Month 6 | Month 6
  Retention rate at 6 months is defined as the percentage of participants remaining on perampanel at 6 months.
Pragmatic Seizure-free Rate at Months 6 and 12 | Months 6 and 12
  Pragmatic seizure-free rate is defined as the percentage of participants (based on all study participants) who are free of all seizures at 6 months (and for the previous 3 months) and at 12 months (and for the previous 6 months).
Completer Seizure-free Rate at Months 6 and 12 | Months 6 and 12
  Completer seizure-free rate is defined as the percentage of participants (based on a subset of study participants who remain on perampanel treatment at 6 and 12 months) who are free of all seizures at 6 months (and for the previous 3 months) and at 12 months (and for the previous 6 months), respectively.
Median Percent Change From Baseline in Seizure Frequency at Months 6 and 12 | Months 6 and 12
  Seizure frequency change will be measured at 6 months (averaged over the previous 3 months) and at 12 months (averaged over the previous 6 months).
50 Percent (%) Responder Rate at Months 6 and 12 | Months 6 and 12
  50% responder rate is defined as the percentage of participants with greater than or equal to (>=) 50% reduction in seizure frequency (averaged over the 3 months before the 6-month visit, and over the 6 months before the12-month visit) relative to baseline.
Seizure Worsening Rate at Months 6 and 12 | Months 6 and 12
  Seizure worsening rate is defined as the percentage of participants with >=10% increase in seizure frequency (averaged over the 3 months before the 6-month visit, and over the 6 months before the 12-month visit) relative to baseline.
Last Dose of Perampanel at Months 6 and 12 | Months 6 and 12
Percentage of Participants by Perampanel Dose Titration Speed | Up to Month 12
Duration of Treatment on Perampanel | Up to Month 12
Percentage of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs),Serious Adverse Events (SAEs), TEAEs Leading to Discontinuation, and TEAEs by Severity | Up to Month 12

CONTACTS AND LOCATIONS:
Locations (36):
- Sydvestjysk Sygehus Esbjerg, Esbjerg, Region Syddanmark, Denmark
- France (8):
  - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - Hôpital Roger Salengro, Lille, Nord
  - Centre de consultations Saint-Jean Bâtiment A, Cagnes-sur-Mer
  - Hopitaux de La Timone, Marseille
  - Hôpital Robert Debré, Paris
  - Centre hospitalier de Pau, Pau
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - CHRU Bretonneau, Tours
- Germany (2):
  - Eisai Trial Site #2, Berlin
  - Eisai Trial Site #1, Ulm
- Italy (9):
  - AORN A Cardarelli, Naples, Campania
  - Azienda Sanitaria Universitaria Integrata di Udine - PO Universitario Santa Maria della Misericordia, Udine, Friuli Venezia Giulia
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - ASST Santi Paolo e Carlo - Azienda Universitaria-Polo Universitario San Paolo, Milan, Lombardy
  - Ospedale di Merano, Merano, Trentino-Alto Adige
  - Ospedale Santa Maria Della Misericordia Di Perugia, Perugia, Umbria
  - Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Policlinico Universitario Campus Biomedico Di Roma, Roma
- Portugal (3):
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Centro Hospitalar Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar de São João, E.P.E., Porto
- Russia (6):
  - Krasnoyarsk State Medical University n.a. V.F. Voyno-Ysenetskiy, Krasnoyarsk
  - City Clinical Hospital #1 n.a. N.I.Pirogov, Moscow
  - Moscow State Medical Stomatological University n.a. A.I. Evdokimov, Moscow
  - Russian National Research Medical University n.a. N.I.Pirogov, Moscow
  - City Neurology Center Sibneuromed LLC, Novosibirsk
  - Regional Treatment and Rehabilitation Center, Tyumen
- Spain (7):
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitari Sagrat Cor Quironsalud, Barcelona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.